CLINICAL TRIAL: NCT06611358
Title: Effect of Kinesio Taping and Exercise Interventions on Pain, Proprioception, Sleep, and Psychological Status in Individuals With Bruxism
Brief Title: The Effects of Kinesio Taping and Exercise Interventions in Individuals With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-4024
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Kinesiology Taping; Bruxism; Exercise
Keywords: kinesiology taping; Bruxism; exercise; temporamandibular disfunction
MeSH Terms: conditions — Bruxism; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology Taping Group (Experimental): Individuals meeting the inclusion criteria will have kinesio tape applied to the temporomandibular joint by a physiotherapist every three days for a duration of two weeks. In addition to the kinesio taping, participants will perform an at-home exercise program prescribed three days a week. This program will include isometric neck exercises (cervical flexion, extension, right and left lateral flexion, right and left rotation, and chin tuck exercises) and temporomandibular joint range of motion exercises (protrusion, retrusion, right and left lateral movement, and mouth opening-closing exercises). As part of the treatment protocol, each movement will be performed in 3 sets of 15 repetitions.
  Interventions: Other: Kinesiology Taping and Exercise
- Conventional Group (Active Comparator): Individuals meeting the inclusion criteria will not receive kinesio taping but will follow the same exercise protocol as the Kinesio Taping + Exercise Group. Participants will perform an exercise program prescribed three days a week, including isometric neck exercises (cervical flexion, extension, right and left lateral flexion, right and left rotation, and chin tuck exercises) and temporomandibular joint range of motion exercises (protrusion, retrusion, right and left lateral movement, and mouth opening-closing exercises). As part of the treatment protocol, each movement will be performed in 3 sets of 15 repetitions.
  Interventions: Other: Convansionel Exercise

INTERVENTIONS:
Other: Kinesiology Taping and Exercise — Individuals meeting the inclusion criteria will receive kinesio taping applied to the temporomandibular joint by a physiotherapist every three days for two weeks. The kinesio tape will be applied along the origin-insertion line with zero tension. In addition to the kinesio taping, participants will follow a exercise program prescribed three days a week. This program will include isometric neck exercises (cervical flexion, extension, right and left lateral flexion, right and left rotation, and chin tuck exercises) and temporomandibular joint range of motion exercises (protrusion, retrusion, right and left lateral movement, and mouth opening-closing exercises). Each movement will be performed as 3 sets of 15 repetitions as part of the treatment protocol
  Arms: Kinesiology Taping Group
Other: Convansionel Exercise — This program will include isometric neck exercises (cervical flexion, extension, right and left lateral flexion, right and left rotation, and chin tuck exercises) and temporomandibular joint range of motion exercises (protrusion, retrusion, right and left lateral movement, and mouth opening-closing exercises). Each movement will be performed as 3 sets of 15 repetitions as part of the treatment protocol.
  Arms: Conventional Group

SUMMARY:
Bruxism is the unconscious act of grinding or clenching the teeth. It leads to hyperactivity of the masticatory muscles due to non-functional mandibular movements, which can result in pain symptoms and is, therefore, a significant factor contributing to changes in the temporomandibular joint. While the beneficial effects of exercise and kinesio taping on temporomandibular dysfunction and bruxism have been validated by various studies in the literature, research investigating their impact on cervical awareness remains quite limited. Hence, the aim of this study is to examine the effects of kinesio taping in addition to exercise on pain, mandibular range of motion, sleep quality, depression levels, and cervical awareness in individuals with bruxism.

DETAILED DESCRIPTION:
Bruxism is a parafunctional or unconscious act of grinding or clenching the teeth. The factors contributing to bruxism are thought to include joint and soft tissue injuries, genetic factors, fatigue, and stress. There is a consensus that the etiology of bruxism is multifactorial and originates from central mechanisms. Bruxism is a common parafunctional activity in the general population, occurring both during sleep and while awake. Daytime bruxism, which is more prevalent in women, affects approximately 20% of the adult population, while sleep bruxism affects around 10%. Overall, the prevalence of bruxism decreases with age, regardless of gender.

The treatment of bruxism aims to raise awareness of oral parafunctional behaviors, alleviate pain, establish a resting position for the temporomandibular joint, improve posture in the head and neck regions, restore muscle strength between affected muscles, and achieve pain-free range of motion. While there is no definitive treatment method, a variety of invasive (acupuncture, injections, surgery, etc.) and non-invasive (exercise, electrical stimulation, manual trigger point stimulation, taping, etc.) approaches are employed. In recent years, reversible non-invasive approaches have gained importance in treatment.

Taping and bandaging have long been part of physiotherapy practices as treatment methods. Kinesio® Tape is a latex-free, thin, cotton-based tape. Developed in Japan 25 years ago, Kinesio® Tape has become widely used in recent years, not only in the United States, Europe, and many other parts of the world but also in our country. The structure, thickness, and weight of the tape are similar to the physical properties of the skin, with a high degree of longitudinal elasticity. The tension levels of the tapes vary depending on the treatment purpose. The primary goal of the Kinesio taping method is to support healing by allowing pain-free movement. In the Kinesio taping method, the tape is applied around or over the muscles as needed to prevent muscle overactivity.

Psychological counseling and exercise are widely used techniques in the treatment of temporomandibular dysfunction (TMD) and have been shown to have positive outcomes in the literature. In a randomized controlled trial by Nimela et al., the efficacy of counseling and masticatory muscle exercises alone was found to be similar to that of stabilization splints in both pain relief and increasing active maximal mouth opening. In a study by Coşkun et al., the addition of kinesio taping to counseling and exercises resulted in significantly greater benefits in both the short and long term. While the beneficial effects of exercise and kinesio taping on TMD and bruxism have been confirmed in various studies, research investigating their impact on cervical awareness is quite limited. Therefore, the aim of this study is to examine the effects of kinesio taping, in addition to exercise, on pain, temporomandibular joint range of motion, sleep quality, depression levels, and cervical awareness in individuals with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Presence of teeth clenching complaints
* Being between the ages of 20 and 50
* No history of major trauma to the Temporamandibular region
* No history of surgical operations on the temporomandibular joint

Exclusion Criteria:

* Individuals with conditions that can cause facial pain, such as sinusitis or trigeminal neuralgia
* Individuals with temporomandibular joint involvement secondary to inflammatory diseases
* Individuals with degenerative problems that restrict neck movements
* Individuals who have received treatment for bruxism in the last 6 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Range of Motion | From enrollment to the end of treatment at 2 weeks
  Maximum mouth opening, protrusion, and lateral movements are jaw motions. Maximum mouth opening is determined by asking the patient to open their mouth as wide as possible and measuring the distance between the maxillary and mandibular incisors.
Pittsburgh Sleep Quality Index | From enrollment to the end of treatment at 2 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported screening and assessment test that provides detailed information on sleep quality, as well as the type and severity of sleep disturbances over the past month. The form consists of 24 questions, from which scores for seven components are obtained: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Of the 24 questions, 19 are self-reported questions. The final five questions, which are answered by the bed partner or roommate, are not included in the scoring and are used only for clinical information. The self-reported questions cover various factors related to sleep quality, including estimates of sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems. The 18 items included in the scoring are grouped into seven component scores. Some components are represented by a single item, while
Beck Depression Inventory | From enrollment to the end of treatment at 2 weeks
  The Beck Depression Inventory (BDI) was developed by Beck, Rush, Shaw, and Emery in 1978 with the aim of measuring somatic, emotional, cognitive, and motivational symptoms commonly observed in depression. The BDI consists of 21 items, each of which has four response options. Each item is scored on a scale from 0 to 3. By summing these scores, a total depression score is obtained. The maximum possible score is 63, with a higher total score indicating a higher level or severity of depression.
Joint Position Sense | From enrollment to the end of treatment at 2 weeks
  The Cervical Joint Position Error Test is used to evaluate cervicocephalic proprioception and neck position sense. This test assesses the ability of the individual to return their head to the original neutral position after maximal rotation in the transverse and sagittal planes. Various devices such as laser pointers, electromagnetic devices, ultrasound-based devices, and electrogoniometers can be used to measure joint position sense error. Among these, using a laser pointer is more practical and easier compared to other methods and is frequently used.
Visual Analogue Scale | From enrollment to the end of treatment at 2 weeks
  The Visual Analog Scale (VAS) consists of a pain level marked by the individual on a plane with a vertical line indicating the pain they are currently experiencing. The pain is rated as 0: no pain at all to 10: the most severe pain imaginable; Scoring is based on measuring the vertical mark made by the participant on the plane using a ruler.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University, Istanbul, Beykoz
  - Istanbul Medipol University, Istanbul

IPD SHARING:
Plan to Share IPD: No